CLINICAL TRIAL: NCT02098187
Title: Pilot 1B Study-Pharmacokinetics of MP-3180 and Use of Noninvasive Fluorescence Detection Device in Healthy Volunteers
Brief Title: Pharmacokinetics of MP-3180 and Use of Noninvasive Fluorescence Detection Device in Healthy Volunteers
Acronym: ORFM-1B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediBeacon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ORFM-1B
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Glomerular Filtration Rate; Acute Kidney Injury
Keywords: Glomerular Filtration Rate; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Below target dose MP-3180 (Active Comparator): 0.5 µmol/kg (0.186 mg/kg) dose of MP-3180 by IV one time over 2 minutes.
  Interventions: Drug: Below target dose MP-3180; Device: ORFM prototype; Other: Iohexol comparator
- 2 times above target dose MP-3180 (Active Comparator): 2 µmol/kg (0.744 mg/kg) dose of MP-3180 by IV one time over 2 minutes.
  Interventions: Drug: 2 times above target dose MP-3180; Device: ORFM prototype; Other: Iohexol comparator
- 4 times above target dose MP-3180 (Active Comparator): 4 µmol/kg (1.488 mg/kg) dose of MP-3180 by IV one time over 2 minutes.
  Interventions: Drug: 4 times above target dose MP-3180; Device: ORFM prototype; Other: Iohexol comparator
- At target dose MP-3180 (Active Comparator): 1 µmol/kg (0.186 mg/kg) dose of MP-3180 by IV one time over 2 minutes.
  Interventions: Drug: At target dose MP-3180; Device: ORFM prototype; Other: Iohexol comparator

INTERVENTIONS:
Drug: Below target dose MP-3180 — MP-3180 0.5 µmol/kg (0.186 mg/kg) dose (fluorescent tracer agent) was administered by IV injection over 2 minutes, followed by a 10 mL saline flush IV over 2 minutes.
  Arms: Below target dose MP-3180
Drug: At target dose MP-3180 — MP-3180 1 µmol/kg (0.186 mg/kg) dose (fluorescent tracer agent) was administered by IV injection over 2 minutes, followed by a 10 mL saline flush IV over 2 minutes.
  Arms: At target dose MP-3180
Drug: 2 times above target dose MP-3180 — MP-3180 2 µmol/kg (0.744 mg/kg) dose (fluorescent tracer agent) was administered by IV injection over 2 minutes, followed by a 10 mL saline flush IV over 2 minutes.
  Arms: 2 times above target dose MP-3180
Drug: 4 times above target dose MP-3180 — MP-3180 4 µmol/kg (1.488 mg/kg) dose (fluorescent tracer agent) was administered by IV injection over 2 minutes, followed by a 10 mL saline flush IV over 2 minutes.
  Arms: 4 times above target dose MP-3180
Device: ORFM prototype — The Optical Renal Function Monitor (ORFM) investigational device noninvasively monitors fluorescent light emission from an exogenous tracer agent over time. Prior to administration of MP-3180 and iohexol, ORFM sensor probes were affixed to each of the participants via standard adhesive pads to four locations: forehead, sternum, upper inner arm, side trunk. The administration of the MP-3180 infusion and iohexol infusion occurred at least 15 minutes after the start of the data acquisition software.
Other: Iohexol comparator — Iohexol (Omnipaque 300, 5 mL) (comparator agent) was administered by IV injection over 2 minutes after MP-3180 injection, followed by a 10 mL saline flush IV over 2 minutes.

SUMMARY:
The purpose of this early feasibility study was to investigate the pharmacokinetics of MP-3180 administered in rising doses and to evaluate the use of the Optical Renal Function Monitor (ORFM), an investigational noninvasive fluorescence detection device.

DETAILED DESCRIPTION:
This was an open-label, rising single-dose study to investigate the pharmacokinetics of the investigational agent, MP-3180, and to evaluate the use of the Optical Renal Function Monitor (ORFM), an investigational noninvasive fluorescence detection device. Single-dose pharmacokinetics at four dose levels were evaluated following the administration of a single, intravenous dose of MP-3180. Iohexol was also administered followed by saline. Prior to administration of MP-3180 and iohexol, ORFM sensor probes were affixed to four locations on the body of each participant. The noninvasive fluorescent signal from MP-3180 was measured using the ORFM investigational device continuously for approximately four hours post MP-3180 administration. For the determination of the pharmacokinetic disposition of MP-3180 and iohexol, blood samples were collected from each participant provided the individual completed all blood collections in the study. The pharmacokinetics of MP-3180 and iohexol were assessed by statistical comparison of pharmacokinetic parameters derived from plasma concentration-time curves and urine recovery data.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 22 years of age or older
2. Sex: Males and not of childbearing potential females
3. Capable of informed consent
4. Weight restrictions:

   1. at least 50 kg (110 lbs) for men
   2. at least 48 kg (106 lbs) for women
   3. all participants will have a Body Mass Index (BMI) less than or equal to 33 but greater than or equal to 19
5. All participants should be judged by the Principal Investigator or Medical Sub-Investigator physician as normal and healthy during a pre-study medical evaluation performed within 28 days of the initial dose of study medication

Exclusion Criteria:

1. Institutionalized participants will not be used
2. History of any significant cardiovascular disease, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic (including any history of seizure disorder), psychological, musculoskeletal disease or malignancies unless deemed not clinically significant by the Principal Investigator or Medical Sub-Investigator.
3. Donation or loss of blood or plasma: 50 mL to 499 mL within 30 days prior to the initial dose of the study medication; or more than 499 mL within 56 days prior to the initial dose of study medication.
4. Intolerance to venipuncture.
5. Participants who have received an investigational drug within 30 days prior to the initial dose of study medication.
6. History of drug and/or alcohol abuse within the past year, unless currently enrolled in an abstinence program.
7. History of allergy or hypersensitivity to MP-3180 or iohexol, or other related products, or any of the inactive ingredients.
8. History of skin sensitivity to adhesives (e.g. Band-Aids, surgical tape).
9. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Principal Investigator or Medical Sub-Investigator, could contraindicate the participant's participation in this study.
10. History of allergy or hypersensitivity to iodine containing contrast media or drugs.
11. Acute illness at the time of either the pre-study medical evaluation or dosing.
12. Social Habits:

    1. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
    2. Ingestion of any vitamins or herbal supplement within 7 days prior to the initial dose of study medication.
    3. Any significant change in dietary or exercise habits within the 48 hours prior to the initial dose of study medication.
13. Medications:

    a. Use of any prescription or over-the-counter (OTC) medications within the 7 days prior to the initial dose of study medication.
14. Not within normal limits or clinically significant for lab testing; serum chemistries, hematology, urinalysis.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Total plasma clearance of MP-3180 and iohexol | Pre-dose and 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. Total plasma clearance (the volume of plasma cleared of the drug over time) was calculated as: Clp = Dose/ AUC∞.
Renal clearance of MP-3180 and iohexol | 60, 120, 240, 360, 600 and 720 minutes post-dose
  Urine samples were collected pre-dose (time 0) and 5 mL urine samples were collected each time the subject voided.
  The total volume of urine excreted was recorded until 12 hours post-dose, and analyzed using validated analytical methods. Renal clearance (the volume of plasma cleared of the drug by the kidneys over time) was calculated as: CLr
  = Ae/ AUClast, where Ae is the cumulative amount of analyte excreted in urine over the sampling interval.
Maximum Plasma Concentration (Cmax) for MP-3180 and iohexol | Pre-dose and 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. Maximum plasma concentration (Cmax; measured in ng/mL) was directly determined from the concentration-time data.
Time to Maximum Plasma Concentration (Tmax) for MP-3180 and iohexol | Pre-dose and 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The time to maximum plasma concentration (Tmax; measured in hours) was directly determined from the concentration-time data.
The terminal rate constant for MP-3180 and iohexol | Pre-dose and 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The terminal rate constant (λz) was determined by linear regression of the terminal linear phase of the log plasma concentration-time profile.
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration for MP-3180 and iohexol | Pre-dose and 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The area under the plasma concentration-time curve (ng*hr/mL) was estimated from time 0 to the last measurable concentration using noncompartmental analyses.
Area under the plasma concentration-time curve from time zero to infinity for MP-3180 and iohexol | Pre-dose and 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The area under the plasma concentration-time curve (ng*hr/mL) from time 0 to infinity was calculated as: AUC∞ = AUClast + LQC/λz where LQC is the predicted concentration (based on the terminal regression) at the time of the last measurable concentration.
The elimination half-life of MP-3180 and iohexol | Pre-dose and 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The elimination half-life (the time required for the concentration of the drug to reach half of its original value) was calculated as t1/2 λz= ln(2)/ λz.

SECONDARY OUTCOMES:
Incidence of adverse events | 1, 3, and 8 hours after dosing, and within 2 weeks after the final study dose
  An adverse event (AE) was defined as any untoward medical occurrence in a study subject after study drug administration and that did not necessarily have a causal relationship with this treatment.
Number of laboratory values that fall outside of pre-specified normal ranges | Pre-dose and within 2 weeks after the final study dose
  Blood samples were collected and analyzed for hematology and clinical chemistry. Out of range values were documented.

OTHER OUTCOMES:
Correlation between MP-3180 fluorescence intensity and MP-3180 concentration in plasma | Pre-dose and 5, 10, 15, 30, 45, 60, 90, 120, 180, 240, 300, 360, 480 and 720 minutes post-dose
  Blood samples were collected and analyzed using validated analytical methods. The fluorescence intensity at the time of the blood sampling was compared to plasma concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B. Dorshow, Ph.D., Study Director — MediBeacon, LLC
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No